CLINICAL TRIAL: NCT02765906
Title: Comparing Different Methods of Patient Education on Preeclampsia: A Randomized Controlled Trial
Brief Title: Comparing Different Methods of Patient Education on Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-0116
Record Dates: First submitted 2016-05-05; First posted 2016-05-09 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Preeclampsia; Anxiety; Hypertension; Pregnancy; Eclampsia; HELLP
Keywords: video; educational tool; preeclampsia; hypertension; pregnancy; patient education; graphic card; eclampsia; HELLP; anxiety; anxiety assessment; STAI 6
MeSH Terms: conditions — Pre-Eclampsia; Anxiety Disorders; Hypertension; Eclampsia | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No intervention (No Intervention): No additional education
- Graphic card (Experimental): Education with graphic card
  Interventions: Other: Graphic card
- Video (Experimental): Education with video
  Interventions: Other: Video

INTERVENTIONS:
Other: Graphic card — A randomized controlled trial comparing patient education on preeclampsia with a graphic card vs. patient education with a written pamphlet vs. no patient education showed that patient education improved significantly when patients were provided with a graphic card depicting signs and symptoms of preeclampsia and that this improvement occurred regardless of health literacy score (You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. American Journal of Obstetrics & Gynecology. 2012;206:431.e1-431.e5.). The graphic card is now available on the Preeclampsia Foundation's website (http://www.preeclampsia.org/market-place/educational-illustrated-signs-symptoms-pad-detail).
  Other Names: Preeclampsia graphic card
  Arms: Graphic card
Other: Video — This an informational video available on the Preeclampsia Foundation's website (http://www.preeclampsia.org/component/allvideoshare/video/featured/7-symptoms-every-pregnant-woman-should-know?Itemid=479). The effectiveness of this video has not yet been tested as an educational tool.
  Other Names: 7 Symptoms Every Pregnant Woman Should Know
  Arms: Video

SUMMARY:
Preeclampsia is a life-threatening condition unique to pregnancy which occurs in 5-8% of all pregnancies. It contributes to a large proportion of maternal mortality worldwide and these deaths largely result from delayed diagnosis.

A number of studies have shown that patient knowledge about preeclampsia is poor and that patient education can improve patient awareness. The investigators would like to find out what type of patient education is most effective. The investigators propose a three arm randomized controlled trial (RCT) where the first arm will receive a graphic card depicting signs and symptoms of preeclampsia, the second arm will watch an educational video on preeclampsia, and the third arm will have no visual form of patient education; they will be exposed only to the counseling they receive with their routine prenatal care. The card and video were both developed by the Preeclampsia Foundation and in a prior RCT the card was shown to be a useful educational intervention. This study would expand on this previous data by comparing the graphic card to an informational video available on the Preeclampsia Foundation's website (http://www.preeclampsia.org/component/allvideoshare/video/featured/7-symptoms-every-pregnant-woman-should-know?Itemid=479). The effectiveness of this video has not yet been tested as an educational tool. Patients in the arm receiving the graphic card for educational intervention will be allowed to keep this card. Primiparous patients seen in the ambulatory prenatal clinic and Maternal Fetal Medicine (MFM) clinic will be enrolled at 18w0d-24w6d gestation. At the time of enrollment baseline preeclampsia knowledge, demographics, and patient anxiety before and after initial exposure to the educational interventions will be assessed. A follow up assessment of knowledge of preeclampsia will be obtained at 32-36 weeks gestation to measure retention of knowledge. Patient medical records will be reviewed for delivery outcomes which will be recorded and compared.

DETAILED DESCRIPTION:
This is a three-arm prospective randomized controlled trial to evaluate patient knowledge of preeclampsia after different forms of education. In the first arm participants will be given a graphic card depicting signs and symptoms of preeclampsia; they will be permitted to keep this card. In the second arm participants will be shown an educational video on preeclampsia. In the third arm participants will have no visual form of patient education; they will be exposed only to the counseling they receive with their routine prenatal care. Participants will be primiparous patients recruited from the prenatal clinic at 18-24 weeks gestation. At time of consent, baseline anxiety assessment with the STAI-6 questionnaire will be obtained followed by a short demographic survey. Participants will be given a short survey on preeclampsia knowledge. They will then be randomized to either preeclampsia education with educational video, graphic card or no visual educational intervention. The participants will be randomized by computer-generated randomization schema (1:1:1). Those randomized to the card will be given a few minutes to review the card. Those randomized to the educational video will watch the video which runs two minutes and 45 seconds. For those randomized to no further intervention, the initial interview will then be over. For the first two arms receiving the graphic card or watching the video, the STAI 6 assessment will be re-administered immediately after the educational intervention and then the interview will be over. Medical record numbers from every participant will be collected for chart review of demographics, preeclampsia risk factors, pregnancy follow up (including triage calls and visits) and delivery outcomes. The participants will be approached again at 32w0d-36w6d gestation to complete a follow up preeclampsia knowledge survey to assess retention of knowledge. This follow-up survey will be collected via phone interview. Participants in the control arm receiving routine prenatal care will also complete a follow up knowledge survey as a control.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women
* English speaking
* Patients at Geisinger Medical Center prenatal clinic
* Patients at Geisinger Medical Center and Forty Fort Maternal Fetal Medicine clinics

Exclusion Criteria:

* Multiparous pregnant women
* Non-English speaking
* Significant hearing loss/disability
* Blind or with severe visual impairment
* Do not have adequate capacity to give consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05; Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Change in percentage of correct responses of preeclampsia knowledge survey score at follow-up assessment | 12-16 weeks
  This survey was previously tested in a study by You et al (You WB, Wolf M, Bailey SC, et al. Factors associated with patient understanding of preeclampsia. Hypertension in pregnancy. 2012;31:341.) and found to have a Cronbach alpha of 0.86. The same survey used in a follow up study by You et al (You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. American Journal of Obstetrics & Gynecology. 2012;206:431.e1-431.e5. )

SECONDARY OUTCOMES:
Change in anxiety level after educational intervention as measured by the STAI 6 | 5 minutes
  The Spielberger State-Trait Anxiety Inventory (STAI) is a reliable and sensitive measure of anxiety at a given moment in time. A shorter form, the STAI-6, was created for efficiency and has been verified as comparable in reliability and validity to the full STAI assessment (Marteau, TM and Beckker, H. The development of a six-item short form of the State Scale of the Spielberger State Trait Anxiety Inventory (STAI). British Journal of Clinical Psychology. 1991: 31: 301-306).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Paglia, MD, PhD, Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger Medical Center: Maternal Fetal Medicine and Prenatal Clinics, Danville, Pennsylvania
  - Geisinger Maternal Fetal Medicine, Forty Fort, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] You WB, Wolf MS, Bailey SC, Grobman WA. Improving patient understanding of preeclampsia: a randomized controlled trial. Am J Obstet Gynecol. 2012 May;206(5):431.e1-5. doi: 10.1016/j.ajog.2012.03.006. Epub 2012 Mar 13. PMID 22542120
- [Background] Firoz T, Sanghvi H, Merialdi M, von Dadelszen P. Pre-eclampsia in low and middle income countries. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):537-48. doi: 10.1016/j.bpobgyn.2011.04.002. Epub 2011 May 17. PMID 21592865
- [Background] Tsigas E, Magee LA. Advocacy organisations as partners in pre-eclampsia progress: patient involvement improves outcomes. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):523-36. doi: 10.1016/j.bpobgyn.2011.03.001. Epub 2011 May 12. PMID 21570359
- [Background] Ogunyemi D, Benae JL, Ukatu C. Is eclampsia preventable? A case control review of consecutive cases from an urban underserved region. South Med J. 2004 May;97(5):440-5. doi: 10.1097/00007611-200405000-00005. PMID 15180017
- [Background] Walker MG, Windrim C, Ellul KN, Kingdom JCP. Web-based education for placental complications of pregnancy. J Obstet Gynaecol Can. 2013 Apr;35(4):334-339. doi: 10.1016/S1701-2163(15)30961-0. PMID 23660041
- [Background] You WB, Wolf M, Bailey SC, Pandit AU, Waite KR, Sobel RM, Grobman W. Factors associated with patient understanding of preeclampsia. Hypertens Pregnancy. 2012;31(3):341-9. doi: 10.3109/10641955.2010.507851. Epub 2010 Sep 22. PMID 20860492
- [Background] Maimburg RD, Vaeth M, Hvidman L, Durr J, Olsen J. Women's worries in first pregnancy: results from a randomised controlled trial. Sex Reprod Healthc. 2013 Dec;4(4):129-31. doi: 10.1016/j.srhc.2013.10.001. Epub 2013 Oct 9. PMID 24216040
- [Background] Muller C, Cameron LD. Trait anxiety, information modality, and responses to communications about prenatal genetic testing. J Behav Med. 2014 Oct;37(5):988-99. doi: 10.1007/s10865-014-9555-8. Epub 2014 Jan 31. PMID 24481564
- [Background] Muthusamy AD, Leuthner S, Gaebler-Uhing C, Hoffmann RG, Li SH, Basir MA. Supplemental written information improves prenatal counseling: a randomized trial. Pediatrics. 2012 May;129(5):e1269-74. doi: 10.1542/peds.2011-1702. Epub 2012 Apr 9. PMID 22492766
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- See also: Related Info — http://www.preeclampsia.org/the-news/videos/video/7-symptoms-every-pregnant-woman-should-know